CLINICAL TRIAL: NCT02083614
Title: The Effect of Clamping the Indwelling Urethral Catheter Before Removal From Patients After Type III Radical Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yao Gong, M.D., First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CIUCGY-1
Record Dates: First submitted 2014-03-08; First posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Gynecologic Cancer

ARMS (2):
- clamping (Experimental): to clamp or release the catheter for 2 days before removal
  Interventions: Procedure: to clamp or release the catheter for 2 days before removal
- no clamping (No Intervention)

INTERVENTIONS:
Procedure: to clamp or release the catheter for 2 days before removal
  Arms: clamping

SUMMARY:
The effect of clamping the indwelling urethral catheter before removal is an unsettled issue in clinical practice. No studies have done before in the patients with gynecologic cancers who received radical hysterectomy. We hypothesized that clamping the catheter would decrease the rate of recatheterization. In addition, the feeling of urination during clamping is correlated with lower rate of recatheterization after removal.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving Piver III radical hysterectomy
* catheterization over 7 days

Exclusion Criteria:

* catheterization shorter than 7 days

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
rate of recatheterization | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fulan Wang, Chongqing, China

REFERENCES:
- [Derived] Ellahi A, Stewart F, Kidd EA, Griffiths R, Fernandez R, Omar MI. Strategies for the removal of short-term indwelling urethral catheters in adults. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD004011. doi: 10.1002/14651858.CD004011.pub4. PMID 34184246